CLINICAL TRIAL: NCT05199454
Title: Role of Adiposomes in Diabetes-Associated Endothelial Dysfunction and Restorative Effects of Exercise and Metabolic Surgery
Brief Title: Role of Adiposomes in Endothelial Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Abeer M. Mohamed, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-1113; 1R01HL161386-01 (NIH)
Record Dates: First submitted 2021-12-19; First posted 2022-01-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Aerobic exercise training for 12 weeks, 3 times per week, 60 minutes per session.
  Interventions: Other: Exercise training
- Control (standards of care) (No Intervention): This arm will receive brochures for healthy lifestyle recommendations. No intervention will be conducted.

INTERVENTIONS:
Other: Exercise training — Aerobic exercise training using a treadmill or a bike for 12 weeks, 3 times per week, 60 minutes per session.
  Arms: Exercise training

SUMMARY:
The development of type II diabetes (T2D) is strongly associated with obesity and both are well-established risk factors for cardiovascular disease. Knowing that vascular dysfunction is an early event in the development of cardiovascular disease in obese diabetic (OB-T2D) patients, The investigators set their long-term goal to define molecular mechanisms of vascular dysfunction and corrective strategies that target these mechanisms such as physical activity and weight loss. The investigators recently discovered that human adipose tissues release extracellular vesicles (adiposomes) that are efficiently captured by endothelial cells. Adiposomes are known to carry bioactive cargos such as proteins and micro RNAs; however, their lipid content has not been studied nor has their ability to transfer their lipid cargo to endothelial cells. In the current application, the investigators propose to investigate the role of adiposomes in communicating the unhealthy milieu, mainly dysregulated lipids, to endothelial cells in OB-T2D subjects. On top of these lipid species that the investigators propose to be carried by adiposomes are glycosphingolipids (GSLs). These lipids originate from the glycosylation of ceramides, a chemical process that is upregulated in the presence of inflammation and high glucose levels. Preliminary findings showed that in endothelial cells, GSL-rich adiposomes disturb plasma membrane structure and subsequently induce endothelial dysfunction. Moreover, the investigators found that preconditioning endothelial cells with high shear stress (which is an exercise mimetic) protected endothelial cells from the detrimental effects induced by adiposomes. Therefore, the central hypothesis is that adipose tissues in OB-T2D patients release GSL-loaded adiposomes that induce vascular endothelial dysfunction. The researchers propose that exercise and weight loss interventions (bariatric surgery) will restore adipose tissue homeostasis, reduce GSL-loaded adiposomes, and subsequently alleviate vascular risk in OB-T2D patients. The investigators will test the hypotheses by pursuing the following aims: aim 1: Investigate the role of GSL-rich adiposomes in the pathogenesis of endothelial dysfunction in OB-T2D adults; aim 2: Test the effectiveness of exercise training in reducing adiposome-mediated effects on vascular function; and aim 3: Examine changes in adiposome/caveolae axis following metabolic surgery and their association with vascular function.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2
* Between ages 18-50 years
* Not pregnant
* Diabetic (Current use of diabetes medication or fasting glucose ≥126 mg/dL)
* Medical clearance to participate in a moderate-intensity exercise program

Exclusion Criteria:

* Pregnant women
* Current smokers
* Currently abusing alcohol or drugs
* Chronic heart, liver, or kidney diseases, autoimmune diseases, or cancer
* Non-English speakers
* History of allergic reactions to lidocaine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation (percent vasodilation) in 60 obese diabetic subjects | 4 years
  Brachial flow-mediated dilation will be measured using ultrasound Alpha 7. For recording, a linear probe will be positioned five centimeters above the left arm's antecubital fossa, and a 1-minute baseline imaging will be recorded. Then, a blood pressure cuff will be put around the right mid-forearm and inflated to 200 to 220 mmHg for 5 minutes. Following cuff deflation (reactive hyperemia), a video grabber will be used to record a 300-second video sequence at three frames per second for offline measurement. The greatest brachial artery diameter at baseline will be deducted from the largest mean values obtained following cuff deflation to determine relative flow mediated dilation

SECONDARY OUTCOMES:
Glycosphingolipid content (ng/ml) in adiposomes from 60 obese diabetic subjects | 4 years
  Adiposomes isolated from adipose tissue samples will be examined for their glycosphingolipid content using mass spectrometry and the outcome will be in nanograms per milliliter (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Abeer M Mohamed, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No